CLINICAL TRIAL: NCT06471127
Title: Genetic and MRI Biomarkers of Neuroplasticity Predict Aphasia Recovery and Phenotypes
Brief Title: Neuroplasticity Biomarkers in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-1101; 1K23DC021744 (NIH); A481800 (Other: UW Madison); L&S/COMMUN SCI & DISORDERS (Other: UW Madison); Protocol Version 9/26/2025 (Other: UW Madison)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Aphasia; Language; Stroke
MeSH Terms: conditions — Aphasia; Language; Stroke

STUDY DESIGN:
Intervention Model Description: Translational. This protocol 1) tests neural mechanisms of connectivity and reorganization that support post-stroke language recovery and 2) determines biomarkers predictive of language impairments to improve prognostics for persons with aphasia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental word-learning task for aphasia (Experimental): The word learning task includes 210 trials across 7 learning blocks (30 trials/block). Each trial features two novel objects (target and foil) on the screen, with an audio recording naming one object. Subjects must quickly and accurately identify the named object. Correct responses are rewarded with a happy face, and incorrect ones with a sad face. The target object's position is counter-balanced, and trial order is randomized for each subject. Short pauses occur every 60 trials to reduce fatigue. After 7 learning blocks, feedback is discontinued, and an immediate test block assesses word-referent recognition. A week later, a second test block, with the same instructions, measures retained learning. Each test block consists of 30 randomized trials without feedback.
  Interventions: Behavioral: Pseudoword learning paradigm task

INTERVENTIONS:
Behavioral: Pseudoword learning paradigm task — Pseudoword learning is an experimental learning task by which participants view two novel objects (a target and a foil) and simultaneously hear an audio recording of the pseudoword name of one of the two objects. Participants must choose (via mouse click) which object corresponds to the word presented, immediately after which feedback is provided.

SUMMARY:
Patients with stroke frequently suffer from aphasia, a disorder of expressive and/or receptive language, that can lead to serious health consequences, including social isolation, depression, reduced quality of life, and increased caregiver burden. Aphasia recovery varies greatly between individuals, and likely relies upon the capacity for neuroplasticity, both at a systems level of reorganized brain networks and a molecular level of neuronal repair and plasticity. The proposed work will evaluate genetic and neural network biological markers of neuroplasticity associated with variability in aphasia, with a future goal to improve prognostics and identify therapeutic targets to reduce the long-term burdens of aphasia.

DETAILED DESCRIPTION:
Aphasia is an acquired neurologic language disorder that is among the most challenging long-term disabilities for stroke survivors, often leading to social isolation and reduced quality of life. Recovery from aphasia relies on plasticity in residual brain networks. However, neuroplasticity varies substantially across individuals, making the presence, severity, and phenotype of language impairments challenging to predict. A vital step toward post-stroke precision medicine is identifying neuroplasticity-related biological markers that can improve prognostic models and targeted neurorehabilitation therapies for people with aphasia. The proposed research will test the central hypothesis that individual differences in neuroplasticity, measured through genetic polymorphisms and longitudinal neuroimaging connectivity biomarkers, will account for significant variance in post-stroke aphasia recovery. This 5-year project will include three specific aims. Aim 1 is to index spontaneous recovery by determining relationships between genetic biomarkers of plasticity, longitudinal neural network connectivity, and changes in language during sub-acute to chronic stroke recovery. Aim 2 is to identify genetic and MRI biomarkers predictive of chronic post-stroke aphasia severity and phenotypes. Aim 3 is to characterize genetic and MRI biomarkers associated with verbal learning variability in chronic aphasia. These data will support the development of a larger, multi-site R01 study to examine interactions between multiple biomarkers of neuroplasticity that inform longitudinal aphasia prognostics and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 40-90
2. Right-handed (prior to stroke)
3. Proficient English speakers
4. History of a single ischemic stroke in the middle cerebral artery territory that is lateralized to the left or right (Aim 1) cerebral hemisphere.
5. Presence of aphasia (Aims 2-3)
6. Capacity to understand the nature of the study and provide informed consent
7. Acute or subacute stroke at the time of Aim 1 enrollment; Stroke #12 months old (chronic) at the time of Aims 2-3 enrollment
8. Medically stable

Exclusion Criteria:

1. History of significant medical or neurological disorder (other than stroke)
2. History of significant or poorly controlled psychiatric disorders
3. Current abuse of alcohol or drugs, prescription or otherwise
4. Clinically significant and uncorrected vision or hearing loss
5. Anything other than standard of care stroke treatment such as Plavix, aspirin (81-300 mg daily), beta-blockers, diabetes medications or choles- terol-lowering agents, thrombolytics (e.g., tPA), anticoagulation agents such as Heparin, Warfarin/Coumadin

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Aphasia presence/severity | 3 months, 6 months, 1 year post-stroke
  The primary outcome measure for Aim 1 will be overall aphasia severity. Severity across language domains will be measured by Western Aphasia Battery-Revised Aphasia Quotient (AQ). AQ scores range from 0-100 and rate severity as follows: 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76+ is mild.
Semantic processing | At least 1 year post-stroke
  A primary outcome measure for Aim 2 will be semantic versus phonological processing ability. Semantic processing will be measured by the three pictures version of the Pyramids and Palm Trees Test (PPT) and Psycholinguistic Assessments of Language Processing in Aphasia (PALPA) 51: Word Semantic Association, and semantic weights will be calculated from Philadelphia Naming Test (PNT).
  PPT ranges from 0-52, with higher scores indicating a better ability to retrieve item names from semantic memory.
  PALPA 51 ranges from 0 to 40, with each correct semantic association earning one point.
  PNT semantic weights refer to the measure of the semantic relatedness of the words used in the test.
Phonological processing | At least 1 year post-stroke
  A primary outcome measure for Aim 2 will be semantic versus phonological processing ability. Phonological processing will be measured by PALPA 1: Same-Different Discrimination Using Nonword Minimal Pairs as a measure of input phonology and phonological weights will be calculated from Philadelphia Naming Test (PNT).
  PALPA 1 range is 0 to 40, with higher scores indicating greater accuracy. PNT phonological weights refer to the measure of the phonologic relatedness of the words used in the test.
Noun processing | At least 1 year post-stroke
  A primary outcome measure for Aim 2 will be noun versus verb processing ability. Noun processing will be measured by Object and Action Naming Battery (OANB) to assess production and Psycholinguistic Assessments of Language Processing in Aphasia (PALPA) 47 to assess comprehension.
  PALPA 47 range is from 0 to 40, with higher scores indicating greater accuracy. OANB object naming range is 0 to 162, with higher scores indicating greater accuracy.
Verb processing | At least 1 year post-stroke
  A primary outcome measure for Aim 2 will be noun versus verb processing ability. Verb processing will be measured by Object and Action Naming to assess production and Northwestern Assessment of Verbs and Sentences (NAVS) Verb Comprehension Test.
  NAVS Verb Comprehension range is 0-22, with higher scores indicating greater accuracy.
  OANB action naming range is 0 to 100, with higher scores indicating greater accuracy.
Pseudoword learning | At least 1 year post-stroke
  A primary outcome measure for Aim 3 will be pseudoword learning, with scores for immediate recognition and delayed recognition ability. This experimental paradigm has been implemented in patients with aphasia by Penaloza and colleagues from the Ancient Farming Equipment Paradigm.
  This assessment is measured in proportion of correction responses, range 0-100%, with higher scores indicating greater accuracy.
Verbal learning | At least 1 year post-stroke
  A primary outcome measure for Aim 3 will be verbal learning, which will be measured by the standardized assessment of Hopkins Verbal Learning Test. Immediate recall is range 0-36 and delayed recall is range 0-12. Higher scores indicate more words recalled. Recognition is range 0-12, with higher scores indicating better ability to correctly identify previously learned information among distractors.

SECONDARY OUTCOMES:
Aphasia Communication Outcome Measure (ACOM) Score | 1 year post-stroke
  The ACOM is a patient-reported measure of communicative effectiveness for persons with aphasia. A final T-score will be scaled such that the mean is 50 and the standard deviation is 10. Higher scores indicate better communicative functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Haley Dresang, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No